CLINICAL TRIAL: NCT06129643
Title: Post-operative Pain After Laser Root Canal Treatment of Necrotic Teeth With Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Post-operative Pain After Laser Root Canal Treatment of Necrotic Teeth With Apical Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Zakaria Fahim, assistant lecturer, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec ID 041909
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pulp Necroses; Apical Periodontitis; Pulp Disease, Dental
Keywords: laser in endodontics; post-operative pain
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis; Dental Pulp Diseases; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional group A (Active Comparator)
  Interventions: Drug: Conventional group
- Dual laser group (Er,Cr:YSGG/Diode) (Experimental)
  Interventions: Device: Dual laser group
- Combined group (EDTA/Diode): (Experimental)
  Interventions: Combination Product: Combined group

INTERVENTIONS:
Drug: Conventional group — conventional disinfection using 2.5% sodium hypochlorite and 17% EDTA
  Other Names: (NaOCl/EDTA)
  Arms: Conventional group A
Device: Dual laser group — Er,Cr:YSGG intracanal laser irradiation to remove smear layer followed by diode laser for disinfection
  Other Names: (Er,Cr:YSGG/Diode)
  Arms: Dual laser group (Er,Cr:YSGG/Diode)
Combination Product: Combined group — 17% EDTA was used to remove smear layer followed by diode laser for disinfection
  Other Names: (EDTA/Diode)
  Arms: Combined group (EDTA/Diode):

SUMMARY:
The aim of this study is to evaluate in vivo the post operative pain after laser root canal treatment in necrotic teeth in an evidence-based clinical trial. The null hypothesis being tested is that there is no difference in post operative pain between conventional irrigation and the two types of lasers used.

Thirty patients are equally divided into 3 separate groups :

* Group A (Conventional): 2.5% NaOCL and 17% EDTA.
* Group B(Dual): saline along with Er,Cr:YSGG laser and diode laser combination
* Group C(Combined): saline along with 17% EDTA and diode laser combination Each patient is given pain scale chart Numeric Rating Scale (NRS) to record his/her pain level before any endodontic treatment. All data will be collected, tabulated, summarized, and statistically analyzed.

DETAILED DESCRIPTION:
Postoperative pain is a common complication following conventional endodontic treatment. According to a systematic review, the frequency of endodontic postoperative pain is between 3% and 58% of patients.Postoperative pain is attributed to chemical, mechanical and microbiological factors.

Residual microorganisms remaining due to the complexity of the root canal system and the limited penetration capability of conventional irrigants are directly responsible for Post operative pain The aim of this study is to evaluate in vivo the post operative pain after laser root canal treatment in necrotic teeth in an evidence-based clinical trial. The null hypothesis being tested is that there is no difference in post operative pain between conventional irrigation and the two types of lasers used.

Thirty patients are equally divided into 3 separate groups :

* Group A (Conventional): 2.5% NaOCL and 17% EDTA.
* Group B(Dual): saline along with Er,Cr:YSGG laser and diode laser combination
* Group C(Combined): saline along with 17% EDTA and diode laser combination Each patient will be given pain scale chart (NRS scale) to record his/her pain level before any endodontic treatment. After disinfection, local anesthetic, tooth isolation, access cavity preparation and final obturation. Patients are asked to mark on a numeric rating scale (NRS) to determine incidence of postoperative pain and rate its intensity at 6, 12, 24, 48, 72 hours, and 7 days after the procedure All data will be collected, tabulated, summarized, and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had asymptomatic, single-rooted maxillary anterior teeth with necrotic pulp and periapical lesion with a periapical index score of 3 or 4
* Patients complaining of no pain and without fistulous tract
* Closed apex.
* Acceptance to participate in the study.

Exclusion Criteria:

* Antibiotic use within the last month, anti-inflammatory analgesic use within the last 5 d, systemic diseases or allergic reactions, calcified canals, root resorption, previous root canal treatment.
* Periodontal diseases, presence of swelling or fistulous tract.
* Vulnerable group including pregnant females, mentally or physically disabled individuals. - Technical difficulties during root canal treatment such as; curved roots, broken files, over instrumentation, overfilling or incomplete filling.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessment | Measure changes in post-operative pain 6 hours after intervention in the three groups using NRS
  Patients will be asked to mark Numeric rating scale (NRS) to determine incidence of postoperative pain and rate its intensity. The NRS consisted of a line anchored by two extremes "No pain" and "the worst pain".
  * Pain level assigned to one of 4 categorical scores:
  * No pain (0), Mild (1-3), Moderate (4-6) and Severe (7-10).
Postoperative pain assessment | Measure changes in post-operative pain 12 hours after intervention in the three groups using NRS
  Patients will be asked to mark Numeric rating scale (NRS) to determine incidence of postoperative pain and rate its intensity. The NRS consisted of a line anchored by two extremes "No pain" and "the worst pain".
  * Pain level assigned to one of 4 categorical scores:
  * No pain (0), Mild (1-3), Moderate (4-6) and Severe (7-10).
Postoperative pain assessment | Measure changes in post-operative pain 24 hours after intervention in the three groups using NRS
  Patients will be asked to mark Numeric rating scale (NRS) to determine incidence of postoperative pain and rate its intensity. The NRS consisted of a line anchored by two extremes "No pain" and "the worst pain".
  * Pain level assigned to one of 4 categorical scores:
  * No pain (0), Mild (1-3), Moderate (4-6) and Severe (7-10).
Postoperative pain assessment | Measure changes in post-operative pain 48 hours after intervention in the three groups using NRS
  Patients will be asked to mark Numeric rating scale (NRS) to determine incidence of postoperative pain and rate its intensity. The NRS consisted of a line anchored by two extremes "No pain" and "the worst pain".
  * Pain level assigned to one of 4 categorical scores:
  * No pain (0), Mild (1-3), Moderate (4-6) and Severe (7-10).
Postoperative pain assessment | Measure changes in post-operative pain 72 hours after intervention in the three groups using NRS
  Patients will be asked to mark Numeric rating scale (NRS) to determine incidence of postoperative pain and rate its intensity. The NRS consisted of a line anchored by two extremes "No pain" and "the worst pain".
  * Pain level assigned to one of 4 categorical scores:
  * No pain (0), Mild (1-3), Moderate (4-6) and Severe (7-10).
Postoperative pain assessment | Measure changes in post-operative pain up to 7 days after intervention in the three groups using NRS
  Patients will be asked to mark Numeric rating scale (NRS) to determine incidence of postoperative pain and rate its intensity. The NRS consisted of a line anchored by two extremes "No pain" and "the worst pain".
  * Pain level assigned to one of 4 categorical scores:
  * No pain (0), Mild (1-3), Moderate (4-6) and Severe (7-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt